CLINICAL TRIAL: NCT02249910
Title: An Open-label, Single Arm, Sequential, Single Centre Trial Investigating the Influence of Oral Semaglutide on Pharmacokinetics of Metformin and Digoxin in Healthy Subjects
Brief Title: Investigating the Influence of Oral Semaglutide on Pharmacokinetics of Metformin and Digoxin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN9924-4145; 2013-004820-12 (EudraCT Number); U1111-1150-0801 (Other: WHO)
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Diabetes; Healthy
MeSH Terms: conditions — Diabetes Mellitus | interventions — semaglutide; Metformin; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Semaglutide (Experimental)
  Interventions: Drug: semaglutide; Drug: metformin; Drug: digoxin; Drug: placebo

INTERVENTIONS:
Drug: semaglutide — Oral administration of 5 mg daily for one week, then escalated to 10 mg daily for one week, followed by escalation to 20 mg daily for 41 days
Drug: metformin — Oral administration of 850 mg twice daily for 3 days followed by 850 mg on day 4, assessed in 3 dosing periods 1) alone, 2) co-administration with SNAC (sodium N-[8-(2-hydroxybenzoyl) amino] caprylate) and 3) co-administration with oral semaglutide.
Drug: digoxin — Oral administration of 0.5 mg single dose, assessed in 3 dosing periods 1) alone, 2) co-administration with SNAC (sodium N-[8-(2-hydroxybenzoyl) amino] caprylate) and 3) co-administration with oral semaglutide.
Drug: placebo — Oral administration of SNAC 300 mg. Will be administered with the morning dose of metformin (1st, 3rd, 5th and 7th dose). On Day 24, a single SNAC dose will be administered with digoxin.

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate the influence of oral semaglutide on pharmacokinetics (the exposure of the trial drug in the body) of metformin and digoxin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18-75 years (both inclusive) at the time of signing inform consent
* Body mass index (BMI) 20.0-29.9 kg/m^2 (both inclusive)
* A good general health based on medical history, physical examination, and results of vital signs, electrocardiogram and laboratory safety tests performed during the screening visit, as judged by the investigator

Exclusion Criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods. Female of child bearing potential must use effective methods of birth control for the duration of the trial and for 5 weeks following last dose. Only highly effective methods of birth control are accepted (i.e., one that results in a less than 1% per year failure rate when used consistently and correctly, such as implants, injectables, combined oral contraceptives, and some intrauterine devices)
* History of Crohn's disease, ulcerative colitis, or other inflammatory bowel disease
* Hypertension (defined as sitting systolic blood pressure above 140 mmHg and/or diastolic blood pressure above 90 mmHg). If white-coat hypertension is suspected at the screening visit a repeated measurement is allowed
* Any blood draw in excess of 25 mL in the past month, or donation of blood or plasma in excess of 400 mL within the 3 months preceding screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2014-09-18 (Actual); Primary Completion 2015-03-06 (Actual); Study Completion 2015-03-06 (Actual)

PRIMARY OUTCOMES:
Area under the metformin plasma concentration-time curve | During a dosing interval (0 to12 hours) at steady state
Area under the digoxin plasma concentration-time curve | From time 0 to infinity after single dose

SECONDARY OUTCOMES:
Maximum observed metformin plasma concentration | During a dosing interval (0 to 12 hours) at steady state
Maximum observed digoxin plasma concentration | 0 to 120 hours after single dose
Maximum observed semaglutide plasma concentration | During a dosing interval (0 to 24 hours) at steady state
Area under the SNAC plasma concentration-time curve | During a dosing interval (0 to 24 hours) at steady state
Number of hypoglycaemic episodes | From the first dosing (Day 1) and until completion of the post treatment follow up visit (Day 118-122)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berlin, Germany

REFERENCES:
- [Background] Baekdal TA, Borregaard J, Hansen CW, Thomsen M, Anderson TW. Effect of Oral Semaglutide on the Pharmacokinetics of Lisinopril, Warfarin, Digoxin, and Metformin in Healthy Subjects. Clin Pharmacokinet. 2019 Sep;58(9):1193-1203. doi: 10.1007/s40262-019-00756-2. PMID 30945118
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com